CLINICAL TRIAL: NCT06693128
Title: Camrelizumab Combined With or Without Apatinib and SOX of Neoadjuvant Treatment for Resectable, Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma: a Prospective, Exploratory II Trial
Brief Title: Camrelizumab Combined With or Without Apatinib and SOX of Neoadjuvant Treatment for Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-019
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — camrelizumab; apatinib; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab and Apatinib and S-1 and Oxaliplatin (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Drug: S-1, Oxaliplatin
- Camrelizumab and S-1 and Oxaliplatin (Experimental)
  Interventions: Drug: Camrelizumab; Drug: S-1, Oxaliplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg
Drug: Apatinib — Apatinib 250mg
  Arms: Camrelizumab and Apatinib and S-1 and Oxaliplatin
Drug: S-1, Oxaliplatin — S-1, Oxaliplatin, q3w

SUMMARY:
This study is a multicenter, randomized, uncontrolled clinical trial to evaluate the efficacy and safety of camrelizumab combined with or without apatinib and SOX of neoadjuvant treatment for resectable locally advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously untreated localized gastric or GEJ adenocarcinoma as defined by T3-4N+M0 (according to AJCC 8th edition) ;
2. Plans to proceed to surgery after completion of neoadjuvant therapy;
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
4. Has adequate organ function.
5. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose, and be willing to use a highly effective method of contraception during the study and for 2 months after the last dose of carrelizumab or 8 weeks after apatinib or 6 months after chemotherapy drugs, whichever is longer.
6. Male subjects whose partners are women of reproductive age should be surgically sterilized or agree to use highly effective methods of contraception during the study and for 2 months after the last administration of carrilizumab or 8 weeks after apatinib or 3 months after chemotherapy drugs, whichever is longer. Sperm donation is not allowed during the study.

Exclusion Criteria:

1. Known HER2 positive;
2. Known peritoneal metastasis or positive peritoneal cytology (CY1P0) or T4b (according to AJCC 8th edition);
3. Previous or concurrent malignancies, except for cured basal cell carcinoma of skin, carcinoma in situ of cervix, and carcinoma in situ of breast;
4. Uncontrolled hypertension ( systolic ≥140 mmHg or diastolic ≥90 mmHg despite antihypertensive therapy)；
5. Known hypersensitivity to any of the study drugs or excipients;
6. Known hereditary or acquired bleeding and thrombotic tendencies (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, etc.);
7. Congenital or acquired immune deficiency (e.g. HIV infected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
  Defined as the percentage of subjects with no residual tumor cells in the primary tumor (Becker Grade 1a)

SECONDARY OUTCOMES:
Major pathological response (MPR) | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
total Pathologic complete response (tpCR) | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
R0 resection rate | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Pathologic Nodal Stage after Neoadjuvant Therapy | Up to 6 weeks after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Event free survival (EFS) | Up to approximately 3 years
Disease-free survival (DFS) | Up to approximately 3 years
Overall survival(OS) | Up to approximately 5 years
AEs | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Zhu, Principal Investigator — Ruijin Hospital; Yantao Tian, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Changhai Hospital, Shanghai
  - Yantai Yuhuangding Hospital, Yantai